CLINICAL TRIAL: NCT04283630
Title: The Combined Effect of Dietary Nitrate and Vitamin C on Endothelial Function, Oxidative Stress Biomarkers, and Blood Lipids
Brief Title: Nitrate and Vitamin C on Vascular Health Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Travis Thomas (Other)
Responsible Party: Sponsor-Investigator, David Travis Thomas, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0412-F3R
Record Dates: First submitted 2020-02-14; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Endothelial Dysfunction
Keywords: Nitrate; Vitamin C; Endothelial function; Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Crossover double blinded crossover study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomization and Dietary supplement Interventions (Active Comparator): The dietary nitrate supplement was provided in the form of commercial beetroot juice (Sport Beet IT shot, Heartbeet Ltd) for all participants, whereas vitamin C and the placebo were provided as supplement capsules. Participants were asked to consume one dose/shot of sport Beet IT (70ml) that delivers on average 300-400mg of inorganic nitrate every day in the morning during the four-week study period, except for the test days and washout weeks. Accordingly, the participant were asked to consume the concentrated beetroot juice with breakfast meals, and then the vitamin C supplement (1000 mg)or placebo at the same time one-hour post beetroot juice supplementation
  Interventions: Dietary Supplement: Dietary nitrate in the form of beetroot juice for all participnats; Dietary Supplement: Nature Made vitamin c 1000 mg
- Placebo (Placebo Comparator): Vitamin C placebo was matched with the active vitamin c capsules in shape, color, and size.
  Interventions: Dietary Supplement: Dietary nitrate in the form of beetroot juice for all participnats; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary nitrate in the form of beetroot juice for all participnats — participants asked to consume dietary nitrate in the form of beet juice everyday in the morning and then one hour later, the vitamin C capsules.
  Other Names: Sport Beet IT shot
Dietary Supplement: Nature Made vitamin c 1000 mg — vitamin C and the placebo were provided as supplement capsules. Participants were asked to consume one dose/shot of sport Beet IT (70ml) that delivers on average 300-400mg of inorganic nitrate every day in the morning during the four-week study period, except for the test days and washout weeks. Accordingly, the participant were asked to consume the daily vitamin C supplement (1000 mg) or placebo one-hour post beetroot juice supplementation.
  Arms: Randomization and Dietary supplement Interventions
Dietary Supplement: Placebo — Vitamin C matched Placebo capsules that made from starch.
  Arms: Placebo

SUMMARY:
The objective of this study is to examine whether the co-administration of dietary nitrate combined with vitamin C for 4 weeks in patients at risk for CVD would yield robust effects on endothelial function using blood measures and a non-invasive technique (Peripheral Artery Tonometry) compared to dietary nitrate supplementation alone.

DETAILED DESCRIPTION:
This is a 10 week randomized, cross-over, double-blinded, placebo-controlled study. This study was designed to compare the magnitude changes in RHI (primary outcome), plasma NO metabolites (nitrate and nitrite), and plasma vitamin C, plasma oxidized LDL, and blood (secondary outcome) following treatment with inorganic nitrate and vitamin C placebo (N) and inorganic nitrate combined with vitamin C (NC). Following baseline testing, eligible subjects were randomized to receive either treatment (N) or treatment (NC) for 4 weeks (period1), and participants were then crossed over to the alternate treatment for another 4 weeks (period 2). There was a 2-week washout at crossover.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 50 and 70 years
* Body mass index (BMI) of 18.5-34.9 kg/m2
* Reactive hyperemia index (RHI) of < or equal to 2
* High cholesterol levels with LDL concentrations (>130 mg/dL)
* Not receiving any lipid lowering therapy.
* Non-smokers

Exclusion Criteria:

* Evidence of overt atherosclerotic disease (i.e., documented medical history of coronary artery disease, peripheral artery disease, cardiovascular disease, and stroke).
* Any surgery or medical history that could confound study results, such as a history of bowel resection, rheumatoid arthritis, inflammatory bowel disease, celiac disease, diabetes, uncontrolled hypertension (systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg), controlled hypertension on clonidine medication.
* Participants were ineligible if they had been diagnosed with the following medical conditions such as active cancer, severe anemia (Hb < 10mg/dL), hepatic or renal disease, heart failure, or finger deformities.
* HIV-positive patients on combination antiretroviral therapy because of potential pharmacokinetic interactions with beetroot juice were excluded.
* Participants were also excluded if they reported taking any form of hormone replacement therapy (estrogens, progesterone, and testosterone), multivitamin supplements that provides >100% of RDA, or any of the following medications that attenuate nitrate conversion to NO: proton pump inhibitors (PPI) and antibiotics.
* Participants who consumed greater than 6 drinks of alcohol (any form) per week, performed structured resistance or aerobic training for more than 1-hour four times per week, or participated in other clinical intervention within the previous 30 days were excluded from the study.
* Eligible subjects were asked to avoid using the mouthwash before and throughout the study duration. In addition, enrolled participants were advised to consume low- vitamin c diet throughout the study. They were provided at the beginning of the study with a list of high vitamin C foods/fortified foods to avoid during the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Change of peripheral endothelial function | Change from baseline endothelial function at 4 weeks of each treatment intervention period
  Non-invasive technique called peripheral artery tonometry reactive hyperemia (PAT-RH)

SECONDARY OUTCOMES:
Change of plasma total nitric oxide (NOx) | Change from baseline plasma NOx at 4 weeks of each treatment intervention period
  Sum of nitric oxide metabolites (nitrite and nitrate) were assessed
Change of blood biomarker of oxidative stress | Change from baseline oxLDL at 4 weeks of each treatment intervention period
  Oxidized low density lipoprotein (oxLDL)
Change of blood lipids | Change from baseline blood lipids at 4 weeks of each treatment intervention period
  Total cholesterol(TC), low density lipoprotein(LDL), triglycerides(TG), and high density lipoprotein (HDL)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basaqr R, Skleres M, Jayswal R, Thomas DT. The effect of dietary nitrate and vitamin C on endothelial function, oxidative stress and blood lipids in untreated hypercholesterolemic subjects: A randomized double-blind crossover study. Clin Nutr. 2021 Apr;40(4):1851-1860. doi: 10.1016/j.clnu.2020.10.012. Epub 2020 Oct 14. PMID 33115598